CLINICAL TRIAL: NCT05681182
Title: A Prospective Pilot Study of the Combination of CardiaMend and Amiodarone for the Prevention of Postoperative Atrial Fibrillation (POAF) in Patients Undergoing Isolated Cardiac Arterial Bypass Grafting or Isolated Valve Surgery (CAMP POAF)
Brief Title: Prevention of Post-OP AFib Using Combination of CardiaMend and Amiodarone
Acronym: CAMP POAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: WakeMed Health and Hospitals (Other)
Collaborators: Helios Cardio Inc. (Industry)
Responsible Party: Principal Investigator, Judson Williams, Principal Investigator, WakeMed Health and Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1937514
Record Dates: First submitted 2022-11-25; First posted 2023-01-12 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Post Operative Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients undergoing isolated cardiac arterial bypass surgery or isolated valve surgery, via complete median sternotomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Other): All patients who are enrolled into the study will receive the treatment. This includes the CardiaMend which should be used according to the Instructions for Use with the exception that device hydration is performed with 3 ampules of amiodarone (150mg/3ml) instead of room temperature saline. For best results, the device should be fixed in place using a continuous or interrupted stitch (approximately 1 stitch per cm) to approximate the edge of the pericardial defect. The closed defect should not put pressure on the underlying structures. A non-absorbable monofilament suture is preferred such as 5-0 or 4-0 prolene. A small edge may be left open for drain placement and a small slit for LIMA in case of CABG
  Interventions: Combination Product: CardiaMend with the Addition of Amiodarone

INTERVENTIONS:
Combination Product: CardiaMend with the Addition of Amiodarone — The CardiaMend patch will be saturated with Amiodarone prior to being sutured into place.

SUMMARY:
The purpose of this study is to evaluate the combination of CardiaMend, with the addition of amiodarone in the prevention of postoperative atrial fibrillation (POAF) in patients undergoing isolated cardiac arterial bypass grafting (CABG) or valve surgery.

DETAILED DESCRIPTION:
This study will investigate CardiaMend, an FDA cleared (K210331) pericardial reconstruction matrix used in combination with amiodarone, an FDA approved antiarrhythmic drug, as a prevention of POAF.

This is a single-center, prospective, pilot study, enrolling adult subjects undergoing isolated cardiac arterial bypass surgery or isolated valve surgery, via complete median sternotomy.

CardiaMend should be used according to the Instructions for Use with the exception that device hydration is performed with 3 ampules of amiodarone (150mg/3ml) instead of room temperature saline. For best results, the device should be fixed in place using a continuous or interrupted stitch (approximately 1 stitch per cm) to approximate the edge of the pericardial defect. The closed defect should not put pressure on the underlying structures. A non-absorbable monofilament suture is preferred such as 5-0 or 4-0 prolene. A small edge may be left open for drain placement and a small slit for LIMA in case of CABG.

Patients will have continuous EKG until discharge. If clinically indicated, patients will receive a monitor for home monitoring per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 20-85 years old.
* Patients able to provide written informed consent, understand, and be willing to comply with study-related procedures.
* Participants who are scheduled to undergo open-chest cardiac surgery via complete median sternotomy. Includes:

  * Coronary artery bypass graft (CABG) or valve repair/replacement, or
  * Inclusionary valve repair/replacement procedures for the primary reason for surgery include: aortic valve repair/replacement, mitral valve repair/replacement.
  * Note: Left atrial appendage (LAA) procedures are allowed if CABG and/or valve repair or replacement is the qualifying surgical procedure, but is not a qualifying surgical procedure on its own.
* In sinus rhythm at the time of office visit and prior EKG (note: continuous EKG monitoring for 48 hours is not required).

Exclusion Criteria:

* Subject unable to give voluntary written informed consent, is unlikely to cooperate or is legally incompetent, including subjects who are institutionalized by court or official order, or in a dependency relationship with, testing center or investigator.
* Any condition which could interfere with the subject's ability to comply with the study.
* Ongoing participation in an interventional clinical study or during the preceding 30 days.
* Female subjects who are pregnant, breastfeeding, were pregnant within the last three months, or are planning to become pregnant during the course of the study.
* Active skin or deep infection at the site of implantation.
* History of chronic wounds or wound-healing disorders.
* Known connective tissue diseases (e.g. Ehlers-Danlos syndrome, Epidermolysis bullosa, Marfan syndrome, Osteogenesis imperfecta).
* Immune-suppressed subjects, immune-deficiency subjects (properly managed diabetes mellitus is not an exclusion criterion).
* Concomitant oral or IV systemic corticosteroid therapy and/or other constant anti-inflammatory therapies.
* The subject has an implantable cardiac device (i.e., cardiac resynchronization therapy devices with and without defibrillator capabilities (CRTs and CRT-Ds), implantable cardioverter-defibrillators (ICD) and pacemakers).
* Known history of atrial fibrillation or paroxysmal atrial fibrillation.
* History of ablation for atrial fibrillation.
* Patients already receiving amiodarone as a treatment for atrial fibrillation or ventricular arrhythmias.
* Disease of the left pleura, previous intervention in the left pleural space, or chest deformity.
* Subjects with end-stage chronic-renal disease / dialysis.
* Subjects with heart failure (BNP>1000), low ejection fraction (<35%), end stage renal disease (on dialysis or creatinine >1.8).
* STS risk >5.5% for 30 day mortality.
* Patients electing to receive an ablative procedure for atrial fibrillation during the index operation.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Post Operative Atrial Fibrillation | Through discharge, an average of 2 weeks
  The patient have continuous ECG monitoring until discharge to evaluate for any evidence of atrial fibrillation or atrial flutter which lasts longer than one hour or if less than one hour, requires medical or procedural intervention

SECONDARY OUTCOMES:
Additional Hospital Time Required Due to Atrial Fibrillation/Flutter | Through discharge, an average of 2 weeks
  Burden of atrial fibrillation as defined by additional treatment regimen, additional time in ICU, complications directly associated with atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Judson B Williams, MD, Principal Investigator — WakeMed Health and Hospitals
Locations (1):
- WakeMed Health and Hospitals, Raleigh, North Carolina, United States

REFERENCES:
- [Result] Rego A, Cheung PC, Harris WJ, Brady KM, Newman J, Still R. Pericardial closure with extracellular matrix scaffold following cardiac surgery associated with a reduction of postoperative complications and 30-day hospital readmissions. J Cardiothorac Surg. 2019 Mar 15;14(1):61. doi: 10.1186/s13019-019-0871-5. PMID 30876459
- [Result] Echahidi N, Pibarot P, O'Hara G, Mathieu P. Mechanisms, prevention, and treatment of atrial fibrillation after cardiac surgery. J Am Coll Cardiol. 2008 Feb 26;51(8):793-801. doi: 10.1016/j.jacc.2007.10.043. PMID 18294562
- [Result] Lowres N, Mulcahy G, Jin K, Gallagher R, Neubeck L, Freedman B. Incidence of postoperative atrial fibrillation recurrence in patients discharged in sinus rhythm after cardiac surgery: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2018 Mar 1;26(3):504-511. doi: 10.1093/icvts/ivx348. PMID 29161419
- [Result] Habbab LM, Chu FV. Intrapericardial Amiodarone for the Prevention of Postoperative Atrial Fibrillation. J Card Surg. 2016 Apr;31(4):253-8. doi: 10.1111/jocs.12700. Epub 2016 Feb 2. PMID 26833498
- [Result] Camm AJ. Safety considerations in the pharmacological management of atrial fibrillation. Int J Cardiol. 2008 Jul 21;127(3):299-306. doi: 10.1016/j.ijcard.2007.11.006. Epub 2008 Jan 8. PMID 18191470
- [Result] Frendl G, Sodickson AC, Chung MK, Waldo AL, Gersh BJ, Tisdale JE, Calkins H, Aranki S, Kaneko T, Cassivi S, Smith SC Jr, Darbar D, Wee JO, Waddell TK, Amar D, Adler D; American Association for Thoracic Surgery. 2014 AATS guidelines for the prevention and management of perioperative atrial fibrillation and flutter for thoracic surgical procedures. J Thorac Cardiovasc Surg. 2014 Sep;148(3):e153-93. doi: 10.1016/j.jtcvs.2014.06.036. Epub 2014 Jun 30. No abstract available. PMID 25129609
- [Result] Beau J, Kulik A. Topical amiodarone to prevent postoperative atrial fibrillation: Need for further study. J Thorac Cardiovasc Surg. 2016 Feb;151(2):600. doi: 10.1016/j.jtcvs.2015.10.007. No abstract available. PMID 26806512